CLINICAL TRIAL: NCT06414434
Title: A Pilot Study of BTX-A51 in Patients With Metastatic and/or Recurrent Liposarcomas Characterized by MDM2 Amplifications, Myxoid Liposarcoma, and CIC-Rearranged Sarcoma
Brief Title: BTX-A51 in Patients With Liposarcoma or CIC-rearranged Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Wagner, MD (Other)
Collaborators: Edgewood Oncology Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Wagner, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-156
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Liposarcoma; Recurrent Liposarcoma; Metastatic Liposarcoma; Unresectable Liposarcoma; MDM2 Gene Amplification; Myxoid Liposarcoma; CIC-Rearranged Sarcoma
Keywords: Liposarcoma; Recurrent Liposarcoma; Metastatic Liposarcoma; Unresectable Liposarcoma; MDM2 Gene Amplification; Myxoid Liposarcoma; CIC-Rearranged Sarcoma
MeSH Terms: conditions — Liposarcoma; Liposarcoma, Myxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BTX-A51 21mg (Experimental): Participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with tumor biopsy.
  * Tumor biopsy at the end of Cycle 1.
  * Radiologic imaging every 2 cycles.
  * Cycle 1 through End of Treatment:
    --Day 1 of 28 day cycle: Predetermined dose of BTX-A51 3x weekly.
  * End of Treatment visit with radiologic imaging.
  * Follow-up: every 3 months for 1 year.
  Interventions: Drug: BTX-A51
- BTX-A51 30mg (Experimental): Participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with tumor biopsy.
  * Tumor biopsy at the end of Cycle 1.
  * Radiologic imaging every 2 cycles.
  * Cycle 1 through End of Treatment:
    --Day 1 of 28 day cycle: Predetermined dose of BTX-A51 3x weekly.
  * End of Treatment visit with radiologic imaging.
  * Follow-up: every 3 months for 1 year.
  Interventions: Drug: BTX-A51

INTERVENTIONS:
Drug: BTX-A51 — Multi-kinase inhibitor, 1.0 mg, 2.0 mg, and 7.0 mg immediate-release capsules, taken orally per protocol.
  Other Names: C32H41ClN6O6S2; (1r,4r)-N 1-(5-chloro-4-(5-(cyclopropylmethyl)-1-methyl-l H pyrazol-3-yl)pyrimidin-2-yl)cyclohexane-l ,4-diamine bis(4-methylbenzenesulfonate),

SUMMARY:
This study is testing two different doses of BTX-A51 to determine if it is safe and tolerable in participants with liposarcoma with MDM2 amplification, myxoid liposarcoma, and CIC-rearranged sarcoma.

The name of the study drug used in this research study is:

-BTX-A51 (a type of kinase inhibitor)

DETAILED DESCRIPTION:
This is a two-cohort, pilot study assessing the safety and preliminary exploration of BTX-A51 at two dose levels in participants with metastatic and/or recurrent liposarcomas characterized by Murine Double Minute Clone 2 (MDM2) amplifications (i.e. de-differentiated and /or well-differentiated liposarcomas), myxoid liposarcoma, and CIC-rearranged sarcomas. BTX-A51 works in a different way from currently approved therapies used to treat liposarcoma by blocking proteins called CK1α and CDK9.

The U.S. Food and Drug Administration (FDA) has not approved BTX-A51 as a treatment for liposarcoma characterized by MDM2 amplifications, myxoid liposarcoma, or CIC-rearranged sarcomas.

The research study procedures include screening for eligibility, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission Tomography (PET) scans, blood tests, and tumor biopsies.

Participants will receive study treatment for as long as there are no serious side effects, and disease does not get worse. Participants will be followed for 1 year after the last dose of BTX-A51.

It is expected that about 24 people will take part in this research study.

Edgewood Oncology is supporting this research study by providing the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have histologically-confirmed metastatic and/or recurrent liposarcoma (limited to the subtypes of well-differentiated and/or dedifferentiated liposarcoma, which are associated with MDM2 amplifications), or myxoid liposarcoma, or CIC-rearranged sarcoma.
* ECOG performance status ≤2
* Adequate organ and marrow function as defined by the following metrics resulted within 7 days of study enrollment:

  * WBC >3000/mm3
  * Platelets >75,000μl
  * ANC >1500μl
  * Hgb >9g/dl
  * Creatinine <1.5 x ULN or measured CrCl of >60ml/m2/1.73 m2
  * Total bilirubin <2 x ULN
  * AST/ALT <3 x ULN
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non- nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as

  ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 11 (Measurement of Effect) for the evaluation of measurable disease.
* Patients must have recovered from toxicity related to prior therapy to grade <=1 (defined by CTCAE v5.0) (except alopecia and neuropathy, or immunotherapy related hypothyroidism)
* As the effect of this study drug on the developing human fetus is not known, women of child-bearing potential and men must agree to use at least 2 methods of contraception (abstinence; hormonal or barrier method of birth control) for the study and at least 2 months after completion.
* Female patient of childbearing potential has a negative serum pregnancy test within 7 days of study enrollment.
* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥18 years
* Patients must have completed all prior anti-cancer treatment for liposarcoma, including radiation, ≥ 14 days prior to registration.

Exclusion Criteria:

* Patient with current evidence of active and uncontrolled infection, NYHA Class III-IV CHF, documented Child's class B-C cirrhosis, or uncontrolled medical disease which in the opinion of the investigator or the sponsor could compromise safety and/or assessment of efficacy.
* Active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative PCR result before enrollment; those who are PCR positive will be excluded.
* Major surgical procedure or open surgical biopsy within 28 days of first dose of study drug
* Active central nervous system (CNS) disease involvement, or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity. Subject with known CNS metastases that are treated and stable (without evidence of CNS toxicity) and are not requiring systemic steroids are allowed to be enrolled.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Myocardial infarction within 12 months of screening
* Use of any other concurrent investigational agents or anticancer agents, excluding hormonal therapy for breast or prostate cancer
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BTX- A51, breastfeeding should be discontinued if the mother is treated with BTX-A51.
* Inability to swallow pills or inadequate GI absorption in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events, with laboratory abnormalities, with dose modifications, delays, interruptions, or premature discontinuation of BTX-A51 due to an adverse event | All AEs will be recorded from the time the subject signs informed consent until 30 days after the last dose of study BTX-A51.
  Safety and tolerability will be monitored through continuous reporting of treatment-emergent and treatment-related adverse events, laboratory abnormalities, and incidence of subjects experiencing dose modifications, delays, interruptions, or premature discontinuation of BTX-A51 due to an adverse event. Toxicities are to be assessed according to the CTCAEv5.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | ORR expected to be observed up to 3 years
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.
1-year Progression-Free Survival (PFS) Rate | 1 year
  1-year PFS is a probability estimated using progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
1-year Overall Survival (OS) | 1 year
  1-year OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wagner, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org